CLINICAL TRIAL: NCT04842032
Title: An Open-label, Multi-center, Single-cohort, Post-marketing Phase 4 Study to Evaluate the Efficacy, Pharmacodynamics, and Safety of the Anti-FGF23 Antibody, KRN23, in Pediatric Chinese Patients With X-linked Hypophosphatemic Rickets/Osteomalacia (XLH)
Brief Title: Study to Assess the Safety, Pharmacokinetics and Efficacy of KRN23 in Pediatric Chinese Patients With XLH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-CN006; CTR20210505 (Other: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: X-linked Hypophosphatemia (XLH)
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN23 (Experimental): KRN23 0.8 mg/kg starting dose, administered Q2W by SC injection up to Week 64. Before KRN23 treatment, all patients will receive oral phosphate and vitamin D analogs for 12 weeks of Run-in period.
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — KRN23 is a sterile clear colourless and preservative free solution supplied in single use 5 mL vials containing 1 mL of KRN23 at a concentration of 30mg/mL
  Other Names: Burosumab; Crysvita

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and efficacy of KRN23 in pediatric Chinese patients with XLH

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese patients, aged 1 to ≤12 years at ICF signature with radiographic evidence of rickets
2. Diagnosis of XLH supported by either of the following:

   * Confirmed PHEX mutation (prior to the study with historic record) in the patient or a directly related family member with approximate X linked inheritance
   * Serum intact FGF23 level ≥30 pg/mL by Kainos assay at Screening
3. Able to receive conventional therapy (oral phosphate and pharmacologic vitamin D)
4. Biochemical findings associated with XLH: Serum phosphorus <3.0 mg/dL (0.97 mmol/L). Serum phosphorus may be re tested (once only) at least 7 days after discontinuation of therapy, if applicable ([see Section 3.1])
5. Serum creatinine within age-adjusted normal range (based on overnight fasting [minimum 4 hours] values collected at Screening)
6. Serum 25(OH)D above or equal to the lower limit of normal (≥16 ng/mL) at Screening. If 25(OH)D levels are below the normal range, 25(OH)D supplementation will be prescribed. Assuming a patient meets all other eligibility requirements, the patient may be re tested for serum 25(OH)D after a minimum of 7 days of treatment
7. Willing to provide access to prior medical records for the collection of historical growth and radiographic data and disease history
8. Written or verbal assent (as appropriate for the patient and region) by the patient and written informed consent by legally authorized representatives provided after the nature of the study has been explained, and prior to any research-related procedures
9. Be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments, as judged by the investigator or subinvestigator
10. Female patients who have reached menarche must have a negative pregnancy test at Screening and be willing to have additional pregnancy testing during the study. If sexually active, male and female patients must be willing to use an effective method of contraception for the duration of the study and for 12 weeks after the last dose of IP

Exclusion Criteria:

1. Positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibody at Screening
2. Tanner stage 4 or higher through physical examination
3. Height percentile >50% based on country specific norms
4. Use of a pharmacologic vitamin D, its metabolites, or analogs, oral phosphate for treatment of XLH, aluminum hydroxide antacids, acetazolamide, thiazide diuretics, and/or systemic corticosteroids within 7 days prior to Week -14
5. Current or prior use of leuprorelin, triptorelin, goserelin, or other drugs known to delay puberty
6. Use of growth hormone therapy within 12 months before ICF signature
7. Have uncontrolled diabetes mellitus, defined as glycated hemoglobin (HbA1c) >8.5% at Screening
8. Presence of nephrocalcinosis on renal ultrasound Grade 4 based on the following scale:
9. Planned or recommended orthopedic surgery (implantation or removal), including staples, 8 plates, or osteotomy, within the first 40 weeks of the study
10. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age adjusted normal limits (based on overnight fasting [minimum 4 hours] values collected at the Screening)
11. Evidence of hyperparathyroidism (parathyroid hormone [PTH] levels 2.5 × ULN)
12. Use of medication to suppress PTH (e.g., Sensipar®, cinacalcet, calcimimetics) within 2 months prior to ICF signature
13. Presence or history of any condition that, in the view of the investigator or subinvestigator, places the subject at high risk of poor treatment compliance or of not completing the study
14. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
15. History of recurrent infection or predisposition to infection, or of known immunodeficiency
16. Use of therapeutic mAb within 90 days prior to ICF signature or history of allergic or anaphylactic reactions to any mAb
17. Presence or history of any hypersensitivity to KRN23 excipients that, in the judgment of the investigator or subinvestigator, places the patient at increased risk for adverse effects
18. Use of any investigational product or investigational medical device within 30 days prior to ICF signature, or need for the use of any investigational agent prior to completion of all scheduled study assessments
19. Other patients who are considered to be ineligible for the study by the investigator or subinvestigator for reasons other than the above

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (CFB) in mean serum phosphorus level at the end of the dose cycle | Weeks 2, 4, 8, 12, 16, 24, 32, 40, 52, and 64

SECONDARY OUTCOMES:
Change in rickets at Weeks 40 and 64 as examined by the Radiograph Global Impression of Change (RGI-C) global score | Weeks 40 and 64
  Changes in the severity of rickets and bowing were assessed using a disease specific qualitative RGI-C scoring system. The RGI-C is a 7-point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets).
Change in Rickets Severity Score (RSS) total score at Weeks 40 and 64 | Weeks 40 and 64
  The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, lucency, separation, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees (the total score is the sum of the wrist and knee score). Higher scores indicate greater rickets severity.
Change in lower extremity skeletal abnormalities, including genu varum and genu valgus, as determined by the RGI-C long leg score at Weeks 40 and 64 | Weeks 40 and 64
  Changes in the severity of lower extremity skeletal abnormalities, including genu varum and genu valgus, were assessed using a disease specific qualitative RGI-C scoring system. The RGI-C is a 7-point ordinal scale with possible values: +3 = very much better (complete or near complete healing), +2 = much better (substantial healing), +1 = minimally better (i.e., minimal healing), 0 = unchanged, -1 = minimally worse (minimal worsening), -2 = much worse (moderate worsening), -3 = very much worse (severe worsening).
Change in serum phosphorus over time | Weeks 0, 1, 2, 4, 8, 12, 16, 24, 32, 40, 52, 64, and 74
Change in serum 1,25-dihydroxyvitamin D (1,25(OH)2D) over time | Weeks 0, 1, 2, 4, 8, 12, 16, 24, 32, 40, 52, 64, and 74
Change in alkaline phosphatase (ALP) over time | Weeks 0, 1, 2, 4, 8, 12, 16, 24, 32, 40, 52, 64, and 74
Change in urinary phosphorus over time | Weeks 0, 1, 2, 4, 8, 12, 16, 24, 32, 40, 52, 64, and 74
Change in ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR; algorithm method) over time | Weeks 0, 1, 2, 4, 8, 12, 16, 24, 32, 40, 52, 64, and 74
Change in recumbent length/standing height in cm, height for age z scores | Weeks 0, 24, 40 and 64
Change in growth velocity from pre-treatment and post-treatment over time | Weeks 0, 24, 40 and 64
Change in growth velocity z scores from pre-treatment and post-treatment over time | Weeks 0, 24, 40 and 64
Six-minute walking test (6MWT) results to examine walking ability (total distance; patients ≥5 years at the time of signing the ICF only) | Weeks 0, 24, 40 and 64
Six-minute walking test (6MWT) results to examine walking ability (percent of predicted normal; patients ≥5 years at the time of signing the ICF only) | Weeks 0, 24, 40 and 64
Ten-item Short Form Health Survey for Children (SF-10) physical domain scores to examine health-related Quality of Life | Weeks 0, 24, 40 and 64
  The SF-10 is a brief, 10-item, guardian-completed assessment designed to measure the physical and psychosocial functioning of children. The physical functioning (PHS) domain includes 5 questions that assess limitations in physical activities because of health problems. The PHS domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
Ten-item Short Form Health Survey for Children (SF-10) Psychosocial scores to examine health-related Quality of Life | Weeks 0, 24, 40 and 64
  The SF-10 is a brief, 10-item, guardian-completed assessment designed to measure the physical and psychosocial functioning of children. The Psychosocial functioning (PSS) domain includes 5 questions that assess limitations in psychosocial activities because of health problems. The PHS domain score was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
Face Pain Scale-Revised (FPS-R) scores to examine health-related Quality of Life | Weeks 0, 24, 40 and 64
  The FPS-R is a dimensionless 10 point Likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain.
Patient-Reported Outcomes Measurement Information System (PROMIS) scores to examine health-related Quality of Life | Weeks 0, 24, 40 and 64
  The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Pain Interference Domain, decreases indicate less pain, for the Physical Function Mobility Domain, increases indicate greater mobility and for the Fatigue Domain, decreases indicate less fatigue.

OTHER OUTCOMES:
Safety of KRN23 by studying the number, severity and relatedness of Adverse Events (including laboratory and imaging assessments) | Week 0 to Week 76
  Incidence, frequency, and severity of AEs and SAEs, including clinically significant changes in laboratory assessments as well as ECHO, ECG, ultrasound, vital sign, X-Ray images and Anti-KRN23 antibody.
Pharmacokinetics (PK): KRN23 concentrations | Weeks 0, 1, 2, 4, 8, 16, 24, 40, 64, and 74
Change from Week -14 to Baseline in serum phosphorus over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in serum 1,25(OH)2D over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in plasma iPTH over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in serum calcium over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in urinary phosphorus over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in TmP/GFR (algorithm method) over time during Run-in Period | Week -14, -10 and -4
Safety of conventional therapy by studying the number, severity and relatedness of Adverse Events | Week -14 to Week 0
  Incidence, frequency, and severity of AEs and SAEs, including clinically significant changes in laboratory assessments during Run-in period

CONTACTS AND LOCATIONS:
Overall Officials: KRN23 Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing
  - Guangzhou Women and Children Medical Center, Guangzhou
  - Shanghai 6th Hospital, Shanghai
  - Shanghai Xinhua Hopsital, Shanghai
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No